CLINICAL TRIAL: NCT01868555
Title: A Randomised, Double-blind, Single Centre, Placebocontrolled, Parallel Group, Multiple s.c. Dose Trial to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Two SIAC Preparations and Two Insulin 454 (SIBA) Preparations in Healthy Japanese Male Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of Two IDegAsp (One Explorative) Preparations and Two Insulin Degludec (One Explorative) Preparations in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1790
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDegAsp 30 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 30; Drug: placebo
- IDegAsp 45 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 45; Drug: placebo
- insulin degludec (B) (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- insulin degludec (E) (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo

INTERVENTIONS:
Drug: insulin degludec — Administered as once daily subcutaneous (s.c., under the skin) dose per 0.6 nmol/kg body weight for 6 days
  Arms: insulin degludec (B); insulin degludec (E)
Drug: insulin degludec/insulin aspart 30 — Administered as once daily subcutaneous (s.c., under the skin) dose per 0.6 nmol/kg body weight for 6 days
  Arms: IDegAsp 30
Drug: insulin degludec/insulin aspart 45 — Administered as once daily subcutaneous (s.c., under the skin) dose per 0.6 nmol/kg body weight for 6 days
  Arms: IDegAsp 45
Drug: placebo — Administered as once daily subcutaneous (s.c., under the skin) dose per 0.6 nmol/kg body weight for 6 days

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to assess the safety, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of two insulin degludec/insulin aspart (IDegAsp) preparations and two insulin degludec (insulin 454) preparations in healthy Japanese male subjects. IDegAsp 45 (B) and insulin degludec (B) are explorative formulations, not similar to the proposed commercial formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male subjects
* Body mass index (BMI) between 18.0 and 27.0 kg/m^2 (both inclusive)
* Body weight above or equal to 50 kg

Exclusion Criteria:

* The receipt of any investigational drug within 16 weeks prior to this trial (the planned first dosing)
* Any clinical laboratory values deviated from the reference range at the laboratory (except for cases within physiological change) or any abnormal electrocardiogram (ECG) findings at the screening, as judged by the investigator or sub-investigator
* Known or suspected allergy to trial product(s) or related products

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Day 1-6 and 7-28 days after day 6

SECONDARY OUTCOMES:
Area under the serum insulin 454 concentration curve | 0-96 hours after last dosing
Area under the serum insulin aspart concentration curve | 0-6 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com